CLINICAL TRIAL: NCT00963235
Title: A Phase 3, Open-label, Single-Arm Trial to Evaluate the Safety, Tolerability, and Immunogenicity of 3 Doses of 13vPnC Vaccine in HIV-Infected Subjects 18 Years of Age or Older Who Have Been Previously Immunized With 23vPS Vaccine
Brief Title: Safety & Immunogenicity of 13vPnC in HIV-Infected Subjects Aged 18 or Older Who Were Previously Immunized With 23vPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 6115A1-3017; B1851028
Record Dates: First submitted 2009-08-20; First posted 2009-08-21 (Estimated); Results first posted 2013-06-10 (Estimated); Last update posted 2013-06-10 (Estimated); Status verified 2013-04

CONDITIONS: HIV Infections; Pneumococcal Infections
Keywords: vaccine; 13-valent pneumococcal conjugate vaccine; human immunodeficiency virus
MeSH Terms: conditions — HIV Infections; Pneumococcal Infections; Acquired Immunodeficiency Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: 13-valent pneumococcal conjugate vaccine; Procedure: Blood draw

INTERVENTIONS:
Biological: 13-valent pneumococcal conjugate vaccine — Three doses of 13vPnC given 6 months apart.
  Other Names: 13vPnC
Procedure: Blood draw — Six blood draws pre-vaccination and 1 month post-vaccination, doses 1-3.

SUMMARY:
The study will evaluate the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate vaccine (13vPnC) in HIV-infected subjects 18 years of age or older who have been previously immunized with at least one dose of 23-valent pneumococcal polysaccharide vaccine (23vPS). All subjects will receive 3 doses of 13vPnC, with each study vaccine dose given approximately 6 months apart.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 years or older at the time of enrollment.
* All female and male subjects who are biologically capable of having children must agree and commit to the use of a reliable method of birth control from the signing of the informed consent form (ICF) until 3 months after the last dose of investigational product.
* Documented vaccination with 1 or more doses of 23vPS at least 6 months before study enrollment.
* CD4+ T-cell count >= 200 cells/µ, obtained on the most recent 2 occasions within 6 months before the first investigational product vaccination.
* HIV-infected subjects with viral load <50,000 copies/mL, obtained on the most recent 2 occasions within 6 months before the first investigational product vaccination.
* Subject is receiving a stable dose of HAART for at least 6 weeks prior to the first investigational product vaccination, or not currently receiving antiretroviral therapy.
* Subject is expected to be available for the entire study period (approximately 18 months) and can be contacted by telephone.
* Subject must be able to complete an electronic diary (e-diary) and complete all relevant study procedures during study participation.
* Subject is deemed to be eligible for the study on the basis of medical history, physical examination, and clinical judgment. (Note: Subjects with preexisting stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease 6 weeks before investigational product vaccination, are eligible.)

Exclusion Criteria:

* Subjects with active AIDS related illness, including opportunistic infections or malignancy.
* Evidence of current illicit substance and/or alcohol abuse, that in the investigator's opinion, precludes the subject from participating in the study or interferes with the evaluation of the study objectives..
* Receipt of any licensed or experimental pneumococcal conjugate vaccine prior to enrollment.
* Contraindication to vaccination with pneumococcal conjugate vaccine.
* Previous anaphylactic reaction to any vaccine or vaccine-related component.
* History of culture-proven invasive disease caused by Streptococcus pneumoniae within the last year.
* Current anticoagulant therapy or a history of bleeding diathesis or any condition associated with prolonged bleeding time that would contraindicate intramuscular injection. (Note: Use of antiplatelet drugs, such as aspirin and clopidogrel, is permitted.)
* Pregnant or breastfeeding women, as defined by history or positive human chorionic gonadotropin (hCG) urine test. All women of childbearing potential must have a urine pregnancy test.
* History of active hepatitis with elevation in pretreatment aspartate aminotransferase (AST) or alanine aminotransferase (ALT) values >5 times the upper limit of normal within the last 6 months.
* Serious chronic disorder or any other disorder that, in the investigator's opinion, precludes the subject from participating in the study or interferes with the evaluation of the study objectives. (Note: Serious chronic disorders include metastatic malignancy, severe chronic obstructive pulmonary disease requiring supplemental oxygen, end-stage renal disease with or without dialysis, and clinically unstable cardiac disease).
* Any major illness/condition that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in and completion of, the study, or could preclude the evaluation of the subject's response.
* History of splenectomy.
* Receipt of any blood products, including immunoglobulin, within 42 days before investigational product vaccination until the last blood draw for the study (approximately 13 months after the first investigational product vaccination).
* Evidence of dementia or other severe cognitive impairment.
* Subject who is, in the opinion of the investigator, unable to receive a vaccination in the deltoid muscle of either arm because of insufficient muscle mass.
* Participation in another study using investigational product from 28 days before study enrollment until the blood draw at visit 6. Between the blood draw at visit 6 and the 6 month follow-up telephone call (visit 7), use of investigational product must be discussed with the Medical Monitor. (Note: Participation in purely observational studies is acceptable.)
* Residence in a nursing home, long-term care facility, or other institution or requirement of semi-skilled nursing care. An ambulatory resident of a retirement home or village is eligible for the trial.
* Subject who is a direct relative (child, grandchild, parent, or grandparent) of study personnel, or who is study personnel.

Temporary Delay Criteria:

* Current febrile illness (oral temperature of =38.0°C [100.4°F]) or other acute illness within 48 hours before study vaccine administration.
* Currently receiving antibiotic therapy, or has completed a course of antibiotic therapy within 10 days before study vaccine administration.
* Receipt of novel influenza A (H1N1) vaccine within 14 days before investigational product vaccination (seasonal influenza vaccine can be given at any time at the discretion of the investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2009-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- United States (11):
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Aurora, Colorado
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- [Derived] Glesby MJ, Watson W, Brinson C, Greenberg RN, Lalezari JP, Skiest D, Sundaraiyer V, Natuk R, Gurtman A, Scott DA, Emini EA, Gruber WC, Schmoele-Thoma B. Immunogenicity and Safety of 13-Valent Pneumococcal Conjugate Vaccine in HIV-Infected Adults Previously Vaccinated With Pneumococcal Polysaccharide Vaccine. J Infect Dis. 2015 Jul 1;212(1):18-27. doi: 10.1093/infdis/jiu631. Epub 2014 Nov 13. PMID 25395187
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-3017&StudyName=Safety%20%26%20Immunogenicity%20of%2013vPnC%20in%20HIV-Infected%20Subjects%20Aged%2018%20or%20Older%20Who%20Were%20Previously%20Immunized%20with%2023vPS

RESULTS

PARTICIPANT FLOW:
Groups:
- 13vPnC: Participants previously immunized with at least 1 dose of 23-valent pneumococcal polysaccharide vaccine (23vPS) received 3 doses of 0.5 milliliter (mL) of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly, 6 months apart.
Period: Overall Study
Arm/Group | 13vPnC
Started | 331
Vaccinated Dose 1 | 329
Vaccinated Dose 2 | 300
Vaccinated Dose 3 | 279
Completed Dose 3 1-month Blood Draw | 277
Completed | 271
Not Completed | 60
Not completed — Withdrawal by Subject | 22
Not completed — Lost to Follow-up | 14
Not completed — Failed to return | 9
Not completed — Protocol Violation | 7
Not completed — Adverse Event | 5
Not completed — Physician Decision | 2
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Safety population included participants who received at least 1 dose of study vaccine.
Arm/Group | 13vPnC
Number analyzed (Participants) | 329
Age Continuous [Mean (Standard Deviation); unit: years] | 47.3 (9.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 263

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Fold Rise (GMFR) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody From 1 Month After Dose 2 of 13vPnC to 1 Month After Dose 3 of 13vPnC
Description: Geometric mean fold rises (GMFRs) for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from 1 month post-dose 2 to 1 month post-dose 3 were computed using the logarithmically transformed assay results. Confidence interval (CI) for the GMFRs were back transformations of a CI based on the Student t distribution for the logarithmically transformed assay results.
Time Frame: 1 month post-dose 2, 1 month post-dose 3
Population: Evaluable immunogenicity population: eligible participants who were >=18 years of age on the day of first vaccination, received at least 2 doses of 13vPnC in the sequence assigned, had valid and determinate assay results, and had no major protocol violations. N (number of participants analyzed)=participants who were evaluable for this measure.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC
Number analyzed (Participants) | 223
fold rise
  Serotype 1 | 0.94 [0.88 to 1.01]
  Serotype 3 | 1.01 [0.95 to 1.08]
  Serotype 4 | 1.01 [0.94 to 1.08]
  Serotype 5 | 0.99 [0.94 to 1.05]
  Serotype 6A | 1.19 [1.11 to 1.27]
  Serotype 6B | 1.21 [1.13 to 1.31]
  Serotype 7F | 1.07 [1.00 to 1.14]
  Serotype 9V | 1.08 [1.02 to 1.15]
  Serotype 14 | 1.08 [0.99 to 1.17]
  Serotype 18C | 1.09 [1.02 to 1.16]
  Serotype 19A | 1.03 [0.98 to 1.09]
  Serotype 19F | 1.17 [1.08 to 1.27]
  Serotype 23F | 1.25 [1.15 to 1.37]

2. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After Dose 3 of 13vPnC Relative to 1 Month After Dose 2 of 13vPnC
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were presented. GMC (13vPnC) and corresponding 2-sided 95 percent (%) CIs were evaluated. Geometric means (GMs) were calculated using all participants with available data for both post-dose 2 and post-dose 3 blood draws.
Time Frame: 1 month post-dose 2, 1 month post-dose 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | 13vPnC
Number analyzed (Participants) | 223
microgram per milliliter (mcg/mL)
  Serotype 1: Dose 2 | 2.31 [1.97 to 2.72]
  Serotype 1: Dose 3 | 2.18 [1.88 to 2.54]
  Serotype 3: Dose 2 | 0.54 [0.47 to 0.62]
  Serotype 3: Dose 3 | 0.55 [0.47 to 0.63]
  Serotype 4: Dose 2 | 1.62 [1.41 to 1.87]
  Serotype 4: Dose 3 | 1.63 [1.42 to 1.88]
  Serotype 5: Dose 2 | 3.26 [2.79 to 3.80]
  Serotype 5: Dose 3 | 3.23 [2.78 to 3.75]
  Serotype 6A: Dose 2 | 3.86 [3.20 to 4.66]
  Serotype 6A: Dose 3 | 4.60 [3.85 to 5.50]
  Serotype 6B: Dose 2 | 4.49 [3.70 to 5.46]
  Serotype 6B: Dose 3 | 5.45 [4.53 to 6.57]
  Serotype 7F: Dose 2 | 3.40 [2.95 to 3.92]
  Serotype 7F: Dose 3 | 3.62 [3.17 to 4.14]
  Serotype 9V: Dose 2 | 2.95 [2.56 to 3.41]
  Serotype 9V: Dose 3 | 3.20 [2.79 to 3.66]
  Serotype 14: Dose 2 | 7.57 [6.27 to 9.15]
  Serotype 14: Dose 3 | 8.16 [6.87 to 9.69]
  Serotype 18C: Dose 2 | 2.75 [2.33 to 3.24]
  Serotype 18C: Dose 3 | 2.99 [2.56 to 3.50]
  Serotype 19A: Dose 2 | 7.57 [6.54 to 8.76]
  Serotype 19A: Dose 3 | 7.80 [6.82 to 8.93]
  Serotype 19F: Dose 2 | 5.73 [4.73 to 6.95]
  Serotype 19F: Dose 3 | 6.70 [5.61 to 8.01]
  Serotype 23F: Dose 2 | 3.80 [3.17 to 4.57]
  Serotype 23F: Dose 3 | 4.77 [4.01 to 5.67]

3. Secondary Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody 1 Month After Dose 2 of 13vPnC Relative to 1 Month After Dose 1 of 13vPnC
Description: Antibody GMC for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were presented. GMC (13vPnC) and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for both post-dose 1 and post-dose 2 blood draws.
Time Frame: 1 month post-dose 1, 1 month post-dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC
Number analyzed (Participants) | 242
mcg/mL
  Serotype 1: Dose 1 | 2.15 [1.80 to 2.57]
  Serotype 1: Dose 2 | 2.36 [2.03 to 2.75]
  Serotype 3: Dose 1 | 0.48 [0.41 to 0.56]
  Serotype 3: Dose 2 | 0.57 [0.49 to 0.65]
  Serotype 4: Dose 1 | 1.37 [1.15 to 1.64]
  Serotype 4: Dose 2 | 1.64 [1.43 to 1.89]
  Serotype 5: Dose 1 | 2.90 [2.48 to 3.40]
  Serotype 5: Dose 2 | 3.29 [2.83 to 3.81]
  Serotype 6A: Dose 1 | 2.80 [2.28 to 3.43]
  Serotype 6A: Dose 2 | 3.86 [3.23 to 4.62]
  Serotype 6B: Dose 1 | 2.90 [2.36 to 3.57]
  Serotype 6B: Dose 2 | 4.47 [3.72 to 5.38]
  Serotype 7F: Dose 1 | 3.45 [2.91 to 4.11]
  Serotype 7F: Dose 2 | 3.41 [2.99 to 3.90]
  Serotype 9V: Dose 1 | 2.63 [2.25 to 3.07]
  Serotype 9V: Dose 2 | 2.99 [2.62 to 3.42]
  Serotype 14: Dose 1 | 6.18 [4.97 to 7.68]
  Serotype 14: Dose 2 | 7.60 [6.35 to 9.09]
  Serotype 18C: Dose 1 | 2.87 [2.37 to 3.48]
  Serotype 18C: Dose 2 | 2.68 [2.29 to 3.13]
  Serotype 19A: Dose 1 | 6.53 [5.54 to 7.69]
  Serotype 19A: Dose 2 | 7.63 [6.65 to 8.74]
  Serotype 19F: Dose 1 | 2.75 [2.18 to 3.49]
  Serotype 19F: Dose 2 | 5.70 [4.75 to 6.84]
  Serotype 23F: Dose 1 | 2.62 [2.11 to 3.25]
  Serotype 23F: Dose 2 | 3.82 [3.21 to 4.56]

4. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After Dose 3 of 13vPnC Relative to 1 Month After Dose 2 of 13vPnC
Description: Serotype-specific OPA GMTs for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) were determined in the blood samples of all the participants using a microcolony OPA (mcOPA) assay. GMT (13vPnC) and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for both post-dose 2 and post-dose 3 blood draws.
Time Frame: 1 month post-dose 2, 1 month post-dose 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | 13vPnC
Number analyzed (Participants) | 219
titers
  Serotype 1: Dose 2 | 41 [32.6 to 50.9]
  Serotype 1: Dose 3 | 49 [40.1 to 61.0]
  Serotype 3: Dose 2 | 44 [36.9 to 52.4]
  Serotype 3: Dose 3 | 56 [47.5 to 66.3]
  Serotype 4: Dose 2 | 703 [567.6 to 870.5]
  Serotype 4: Dose 3 | 724 [585.2 to 896.6]
  Serotype 5: Dose 2 | 67 [51.9 to 86.1]
  Serotype 5: Dose 3 | 74 [57.6 to 94.2]
  Serotype 6A: Dose 2 | 1780 [1392.7 to 2274.5]
  Serotype 6A: Dose 3 | 2139 [1709.0 to 2678.3]
  Serotype 6B: Dose 2 | 1857 [1509.8 to 2284.3]
  Serotype 6B: Dose 3 | 2447 [2011.9 to 2977.3]
  Serotype 7F: Dose 2 | 942 [778.6 to 1139.6]
  Serotype 7F: Dose 3 | 1041 [846.5 to 1279.4]
  Serotype 9V: Dose 2 | 657 [482.7 to 893.4]
  Serotype 9V: Dose 3 | 922 [696.0 to 1221.7]
  Serotype 14: Dose 2 | 746 [614.8 to 905.8]
  Serotype 14: Dose 3 | 819 [684.7 to 978.8]
  Serotype 18C: Dose 2 | 521 [383.9 to 706.2]
  Serotype 18C: Dose 3 | 692 [516.2 to 927.7]
  Serotype 19A: Dose 2 | 401 [340.2 to 473.0]
  Serotype 19A: Dose 3 | 419 [358.2 to 490.5]
  Serotype 19F: Dose 2 | 269 [202.3 to 357.3]
  Serotype 19F: Dose 3 | 245 [184.2 to 325.8]
  Serotype 23F: Dose 2 | 293 [217.2 to 395.0]
  Serotype 23F: Dose 3 | 393 [295.0 to 522.7]

5. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMTs) 1 Month After Dose 2 of 13vPnC Relative to 1 Month After Dose 1 of 13vPnC
Description: as for outcome 4
Time Frame: 1 month post-dose 1, 1 month post-dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | 13vPnC
Number analyzed (Participants) | 241
titers
  Serotype 1: Dose 1 | 40 [32.2 to 50.2]
  Serotype 1: Dose 2 | 40 [32.6 to 49.7]
  Serotype 3: Dose 1 | 29 [24.0 to 34.9]
  Serotype 3: Dose 2 | 43 [36.4 to 51.4]
  Serotype 4: Dose 1 | 622 [478.8 to 806.9]
  Serotype 4: Dose 2 | 695 [568.1 to 850.7]
  Serotype 5: Dose 1 | 66 [51.2 to 85.7]
  Serotype 5: Dose 2 | 65 [50.8 to 82.1]
  Serotype 6A: Dose 1 | 976 [710.3 to 1342.0]
  Serotype 6A: Dose 2 | 1687 [1317.2 to 2159.5]
  Serotype 6B: Dose 1 | 1088 [806.0 to 1468.4]
  Serotype 6B: Dose 2 | 1789 [1443.4 to 2216.8]
  Serotype 7F: Dose 1 | 786 [606.6 to 1018.0]
  Serotype 7F: Dose 2 | 927 [763.6 to 1125.2]
  Serotype 9V: Dose 1 | 423 [300.6 to 594.1]
  Serotype 9V: Dose 2 | 695 [518.3 to 932.0]
  Serotype 14: Dose 1 | 640 [509.2 to 805.7]
  Serotype 14: Dose 2 | 723 [602.4 to 867.2]
  Serotype 18C: Dose 1 | 475 [338.5 to 665.5]
  Serotype 18C: Dose 2 | 562 [421.7 to 748.9]
  Serotype 19A: Dose 1 | 299 [239.7 to 372.2]
  Serotype 19A: Dose 2 | 391 [333.2 to 458.6]
  Serotype 19F: Dose 1 | 132 [93.6 to 185.0]
  Serotype 19F: Dose 2 | 247 [189.3 to 322.9]
  Serotype 23F: Dose 1 | 92 [65.6 to 127.9]
  Serotype 23F: Dose 2 | 269 [201.3 to 360.7]

6. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rise (GMFR) From 1 Month After Dose 2 of 13vPnC to 1 Month After Dose 3 of 13vPnC
Description: GMFRs for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from 1 month post-dose 2 to 1 month post-dose 3 were computed using the logarithmically transformed assay results. CI for the GMFRs were back transformations of a CI based on the Student t distribution for the logarithmically transformed assay results.
Time Frame: 1 month post-dose 2, 1 month post-dose 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC
Number analyzed (Participants) | 219
fold rise
  Serotype 1 | 1.2 [1.06 to 1.39]
  Serotype 3 | 1.3 [1.13 to 1.44]
  Serotype 4 | 1.0 [0.90 to 1.18]
  Serotype 5 | 1.1 [0.95 to 1.28]
  Serotype 6A | 1.2 [1.04 to 1.39]
  Serotype 6B | 1.3 [1.16 to 1.50]
  Serotype 7F | 1.1 [0.95 to 1.28]
  Serotype 9V | 1.4 [1.09 to 1.81]
  Serotype 14 | 1.1 [0.97 to 1.24]
  Serotype 18C | 1.3 [1.10 to 1.60]
  Serotype 19A | 1.0 [0.95 to 1.15]
  Serotype 19F | 0.9 [0.76 to 1.09]
  Serotype 23F | 1.3 [1.16 to 1.56]

7. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rise (GMFR) From 1 Month After Dose 1 of 13vPnC to 1 Month After Dose 2 of 13vPnC
Description: GMFRs for the 13 serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from 1 month post-dose 1 to 1 month post-dose 2 were computed using the logarithmically transformed assay results. CI for the GMFRs were back transformations of a CI based on the Student t distribution for the logarithmically transformed assay results.
Time Frame: 1 month post-dose 1, 1 month post-dose 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 13vPnC
Number analyzed (Participants) | 241
fold rise
  Serotype 1 | 1.0 [0.84 to 1.20]
  Serotype 3 | 1.5 [1.29 to 1.73]
  Serotype 4 | 1.1 [0.92 to 1.36]
  Serotype 5 | 1.0 [0.79 to 1.20]
  Serotype 6A | 1.7 [1.39 to 2.15]
  Serotype 6B | 1.6 [1.34 to 2.02]
  Serotype 7F | 1.2 [0.96 to 1.45]
  Serotype 9V | 1.6 [1.26 to 2.14]
  Serotype 14 | 1.1 [0.98 to 1.30]
  Serotype 18C | 1.2 [0.95 to 1.47]
  Serotype 19A | 1.3 [1.15 to 1.50]
  Serotype 19F | 1.9 [1.48 to 2.39]
  Serotype 23F | 2.9 [2.29 to 3.77]

8. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: 13vPnC Dose 1
Description: Specific local reactions were prompted for each day, and reported using an electronic diary. Redness and Swelling scaled as Any (redness present or swelling present); Mild (2.5 to 5.0 centimeters [cm]); Moderate (5.5 to 10.0 cm); Severe (greater than [>] 10 cm). Pain scaled as Any (pain present); Mild (awareness of pain; easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating).
Time Frame: Within 14 days post-dose 1
Population: Safety population:participants who received at least 1 dose of study vaccine. 'N'(number of participants analyzed)=participants whose response was "Yes" for any day or "No" for all days. 'n' = participants whose response was "Yes" for any day or "No" for all days for specified local reaction. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 261
percentage of participants
  Redness: any (n = 162) | 5.6 [2.6 to 10.3]
  Redness: mild (n = 161) | 4.3 [1.8 to 8.8]
  Redness: moderate (n = 158) | 1.3 [0.2 to 4.5]
  Redness: severe (n = 157) | 0.0 [0.0 to 2.3]
  Swelling: any (n = 162) | 6.8 [3.4 to 11.8]
  Swelling: mild (n = 161) | 6.2 [3.0 to 11.1]
  Swelling: moderate (n = 158) | 0.6 [0.0 to 3.5]
  Swelling: severe (n = 158) | 0.6 [0.0 to 3.5]
  Pain: any (n = 260) | 78.8 [73.4 to 83.6]
  Pain: mild (n = 258) | 76.4 [70.7 to 81.4]
  Pain: moderate (n = 173) | 18.5 [13.0 to 25.1]
  Pain: severe (n = 158) | 1.3 [0.2 to 4.5]

9. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: 13vPnC Dose 2
Description: Specific local reactions were prompted for each day, and reported using an electronic diary. Redness and Swelling scaled as Any (redness present or swelling present); Mild (2.5 to 5.0 cm); Moderate (5.5 to 10.0 cm); Severe (>10 cm). Pain scaled as Any (pain present); Mild (awareness of pain; easily tolerated); Moderate (discomfort enough to cause interference with usual activity); Severe (incapacitating).
Time Frame: Within 14 days post-dose 2
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 238
percentage of participants
  Redness: any (n = 122) | 8.2 [4.0 to 14.6]
  Redness: mild (n = 120) | 6.7 [2.9 to 12.7]
  Redness: moderate (n = 117) | 1.7 [0.2 to 6.0]
  Redness: severe (n = 117) | 1.7 [0.2 to 6.0]
  Swelling: any (n = 126) | 12.7 [7.4 to 19.8]
  Swelling: mild (n = 125) | 12.0 [6.9 to 19.0]
  Swelling: moderate (n = 116) | 0.9 [0.0 to 4.7]
  Swelling: severe (n = 117) | 1.7 [0.2 to 6.0]
  Pain: any (n = 237) | 81.4 [75.9 to 86.2]
  Pain: mild (n = 230) | 78.7 [72.8 to 83.8]
  Pain: moderate (n = 150) | 33.3 [25.9 to 41.5]
  Pain: severe (n = 123) | 8.1 [4.0 to 14.4]

10. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Local Reactions: 13vPnC Dose 3
Description: as for outcome 9
Time Frame: Within 14 days post-dose 3
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 205
percentage of participants
  Redness: any (n = 105) | 9.5 [4.7 to 16.8]
  Redness: mild (n = 104) | 8.7 [4.0 to 15.8]
  Redness: moderate (n = 102) | 3.9 [1.1 to 9.7]
  Redness: severe (n = 101) | 1.0 [0.0 to 5.4]
  Swelling: any (n = 107) | 11.2 [5.9 to 18.8]
  Swelling: mild (n = 106) | 8.5 [4.0 to 15.5]
  Swelling: moderate (n = 102) | 3.9 [1.1 to 9.7]
  Swelling: severe (n = 101) | 1.0 [0.0 to 5.4]
  Pain: any (n = 204) | 81.9 [75.9 to 86.9]
  Pain: mild (n = 197) | 80.2 [73.9 to 85.5]
  Pain: moderate (n = 129) | 30.2 [22.5 to 38.9]
  Pain: severe (n = 105) | 5.7 [2.1 to 12.0]

11. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: 13vPnC Dose 1
Description: Specific systemic events (fever greater than or equal to [>=]38 degrees Celsius[C], fatigue, headache, vomiting, diarrhea, new generalized muscle/joint pain and use of medication to treat pain/fever) were prompted for each day, and reported using an electronic diary. Fatigue, headache, new generalized muscle and joint pain were scaled as: Any (symptom present); Mild (no interference with activity); Moderate (some interference); Severe (prevents routine daily activity). Vomiting was scaled as: Any (vomiting present); Mild (1-2 times in 24 hours [hrs]); Moderate (>2 times in 24 hrs); Severe (requires intravenous hydration). Diarrhea was scaled as: Any (diarrhea present); Mild (2-3 loose stools in 24 hrs); Moderate (4-5 loose stools 24 hrs); Severe (>=6 loose stools in 24 hrs). Report of fever >40 degrees C after 13vPnC Dose 1 was confirmed as data entry error.
Time Frame: Within 14 days post-dose 1
Population: Safety population:participants who received at least 1 dose of study vaccine. 'N'(number of participants analyzed)=participants whose response was "Yes" for any day or "No" for all days. 'n' = participants whose response was "Yes" for any day or "No" for all days for specified systemic event. Participants may be represented in more than 1 category.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 276
percentage of participants
  Fever >=38 degrees C (n = 162) | 6.2 [3.0 to 11.1]
  Fever >=38, <38.5 degrees C (n = 160) | 3.8 [1.4 to 8.0]
  Fever >=38.5, <39 degrees C (n = 157) | 1.3 [0.2 to 4.5]
  Fever >=39, =<40 degrees C (n = 159) | 1.3 [0.2 to 4.5]
  Fever >40 degrees C (n = 158) | 0.6 [0.0 to 3.5]
  Fatigue: any (n = 235) | 60.0 [53.4 to 66.3]
  Fatigue: mild (n = 223) | 54.3 [47.5 to 60.9]
  Fatigue: moderate (n = 200) | 37.5 [30.8 to 44.6]
  Fatigue: severe (n = 163) | 6.1 [3.0 to 11.0]
  Headache: any (n = 224) | 61.6 [54.9 to 68.0]
  Headache: mild (n = 216) | 57.4 [50.5 to 64.1]
  Headache: moderate (n = 183) | 31.1 [24.5 to 38.4]
  Headache: severe (n = 160) | 3.1 [1.0 to 7.1]
  Vomiting: any (n = 164) | 11.6 [7.1 to 17.5]
  Vomiting: mild (n = 164) | 11.6 [7.1 to 17.5]
  Vomiting: moderate (n = 157) | 0.0 [0.0 to 2.3]
  Vomiting: severe (n = 157) | 0.0 [0.0 to 2.3]
  Diarrhea: any (n = 193) | 44.0 [36.9 to 51.3]
  Diarrhea: mild (n = 191) | 40.3 [33.3 to 47.6]
  Diarrhea: moderate (n = 166) | 12.7 [8.0 to 18.7]
  Diarrhea: severe (n = 160) | 1.9 [0.4 to 5.4]
  New generalized muscle pain: any (n = 234) | 65.0 [58.5 to 71.1]
  New generalized muscle pain: mild (n = 230) | 60.4 [53.8 to 66.8]
  New generalized muscle pain: moderate (n = 183) | 29.5 [23.0 to 36.7]
  New generalized muscle pain: severe (n = 161) | 3.7 [1.4 to 7.9]
  New generalized joint pain: any (n = 193) | 35.8 [29.0 to 43.0]
  New generalized joint pain: mild (n = 185) | 29.7 [23.2 to 36.9]
  New generalized joint pain: moderate (n = 172) | 19.2 [13.6 to 25.9]
  New generalized joint pain: severe (n = 159) | 1.3 [0.2 to 4.5]
  Use of medication to treat pain (n = 185) | 29.7 [23.2 to 36.9]
  Use of medication to treat fever (n = 173) | 17.3 [12.0 to 23.8]

12. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: 13vPnC Dose 2
Description: Specific systemic events (fever >=38 degrees C, fatigue, headache, vomiting, diarrhea, new generalized muscle/joint pain and use of medication to treat pain/fever) were prompted for each day, and reported using an electronic diary. Fatigue, headache, new generalized muscle and joint pain were scaled as: Any (symptom present); Mild (no interference with activity); Moderate (some interference); Severe (prevents routine daily activity). Vomiting was scaled as: Any (vomiting present); Mild (1-2 times in 24 hrs); Moderate (>2 times in 24 hrs); Severe (requires intravenous hydration). Diarrhea was scaled as: Any (diarrhea present); Mild (2-3 loose stools in 24 hrs); Moderate (4-5 loose stools 24 hrs); Severe (>=6 loose stools in 24 hrs).
Time Frame: Within 14 days post-dose 2
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 229
percentage of participants
  Fever >=38 degrees C (n = 117) | 5.1 [1.9 to 10.8]
  Fever >=38, <38.5 degrees C (n = 116) | 4.3 [1.4 to 9.8]
  Fever >=38.5, <39 degrees C (n = 116) | 0.9 [0.0 to 4.7]
  Fever >=39, =<40 degrees C (n = 115) | 0.0 [0.0 to 3.2]
  Fever >40 degrees C (n = 115) | 0.0 [0.0 to 3.2]
  Fatigue: any (n = 188) | 63.3 [56.0 to 70.2]
  Fatigue: mild (n = 176) | 57.4 [49.7 to 64.8]
  Fatigue: moderate (n = 154) | 38.3 [30.6 to 46.5]
  Fatigue: severe (n = 121) | 7.4 [3.5 to 13.7]
  Headache: any (n = 173) | 56.1 [48.3 to 63.6]
  Headache: mild (n = 165) | 48.5 [40.6 to 56.4]
  Headache: moderate (n = 142) | 31.0 [23.5 to 39.3]
  Headache: severe (n = 117) | 3.4 [0.9 to 8.5]
  Vomiting: any (n = 120) | 7.5 [3.5 to 13.8]
  Vomiting: mild (n = 119) | 6.7 [2.9 to 12.8]
  Vomiting: moderate (n = 116) | 0.9 [0.0 to 4.7]
  Vomiting: severe (n = 115) | 0.0 [0.0 to 3.2]
  Diarrhea: any (n = 155) | 44.5 [36.5 to 52.7]
  Diarrhea: mild (n = 147) | 39.5 [31.5 to 47.8]
  Diarrhea: moderate (n = 130) | 15.4 [9.7 to 22.8]
  Diarrhea: severe (n = 119) | 5.0 [1.9 to 10.7]
  New generalized muscle pain: any (n = 199) | 71.9 [65.1 to 78.0]
  New generalized muscle pain: mild (n = 188) | 66.0 [58.7 to 72.7]
  New generalized muscle pain: moderate (n = 153) | 38.6 [30.8 to 46.8]
  New generalized muscle pain: severe (n = 125) | 10.4 [5.7 to 17.1]
  New generalized joint pain: any (n = 150) | 40.0 [32.1 to 48.3]
  New generalized joint pain: mild (n = 144) | 34.7 [27.0 to 43.1]
  New generalized joint pain: moderate (n = 135) | 21.5 [14.9 to 29.4]
  New generalized joint pain: severe (n = 119) | 3.4 [0.9 to 8.4]
  Use of medication to treat pain (n = 141) | 35.5 [27.6 to 44.0]
  Use of medication to treat fever (n = 127) | 18.9 [12.5 to 26.8]

13. Other Pre Specified Outcome: Percentage of Participants Reporting Pre-Specified Systemic Events: 13vPnC Dose 3
Description: as for outcome 12
Time Frame: Within 14 days post-dose 3
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 13vPnC
Number analyzed (Participants) | 203
percentage of participants
  Fever >=38 degrees C (n = 104) | 7.7 [3.4 to 14.6]
  Fever >=38, <38.5 degrees C (n = 104) | 4.8 [1.6 to 10.9]
  Fever >=38.5, <39 degrees C (n = 101) | 1.0 [0.0 to 5.4]
  Fever >=39, =<40 degrees C (n = 101) | 2.0 [0.2 to 7.0]
  Fever >40 degrees C (n = 101) | 0.0 [0.0 to 3.6]
  Fatigue: any (n = 160) | 56.3 [48.2 to 64.1]
  Fatigue: mild (n = 149) | 48.3 [40.1 to 56.6]
  Fatigue: moderate (n = 132) | 36.4 [28.2 to 45.2]
  Fatigue: severe (n = 105) | 5.7 [2.1 to 12.0]
  Headache: any (n = 137) | 46.7 [38.1 to 55.4]
  Headache: mild (n = 130) | 40.8 [32.2 to 49.7]
  Headache: moderate (n = 118) | 24.6 [17.1 to 33.4]
  Headache: severe (n = 103) | 4.9 [1.6 to 11.0]
  Vomiting: any (n = 109) | 11.0 [5.8 to 18.4]
  Vomiting: mild (n = 107) | 8.4 [3.9 to 15.4]
  Vomiting: moderate (n = 104) | 4.8 [1.6 to 10.9]
  Vomiting: severe (n = 101) | 0.0 [0.0 to 3.6]
  Diarrhea: any (n = 134) | 38.8 [30.5 to 47.6]
  Diarrhea: mild (n = 131) | 35.9 [27.7 to 44.7]
  Diarrhea: moderate (n = 109) | 11.9 [6.5 to 19.5]
  Diarrhea: severe (n = 103) | 1.9 [0.2 to 6.8]
  New generalized muscle pain: any (n = 170) | 65.9 [58.2 to 73.0]
  New generalized muscle pain: mild (n = 155) | 61.3 [53.1 to 69.0]
  New generalized muscle pain: moderate (n = 132) | 31.1 [23.3 to 39.7]
  New generalized muscle pain: severe (n = 110) | 10.0 [5.1 to 17.2]
  New generalized joint pain: any (n = 129) | 31.8 [23.9 to 40.6]
  New generalized joint pain: mild (n = 119) | 26.1 [18.4 to 34.9]
  New generalized joint pain: moderate (n = 120) | 20.0 [13.3 to 28.3]
  New generalized joint pain: severe (n = 106) | 5.7 [2.1 to 11.9]
  Use of medication to treat pain (n = 122) | 32.0 [23.8 to 41.0]
  Use of medication to treat fever (n = 118) | 25.4 [17.9 to 34.3]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs)/serious AEs (SAEs): recorded from signing of informed consent form to completion of study. Participants recorded pre-specified AEs in electronic diary:local reactions; systemic events (up to 14 days after each vaccine dose)
Description: SAEs, AEs were grouped by system organ class and summarized. AEs included AEs collected in electronic diary (local and systemic reactions;systematic assessment), events collected on case report form at each visit (nonsystematic assessment). 1 Participant received Dose 3 but had no safety data available;hence 278 evaluable in after Dose 3 group.
Groups:
- 13vPnC (After Dose 1 and Before Dose 2): Participants who were previously immunized with at least 1 dose of 23-valent pneumococcal polysaccharide vaccine (23vPS), received 1 dose of 0.5 milliliter (mL) of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly and were assessed from 13vPnC Dose 1 to prior to administration of 13vPnC Dose 2.
- 13vPnC (After Dose 2 and Before Dose 3): Participants who were previously immunized with at least 1 dose of 23-valent pneumococcal polysaccharide vaccine (23vPS), received 2 doses of 0.5 milliliter (mL) of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly 6 months apart and were assessed from 13vPnC Dose 2 prior to administration of 13vPnC Dose 3.
- 13vPnC (After Dose 3 and Before Dose 3 Blood Draw): Participants who were previously immunized with at least 1 dose of 23-valent pneumococcal polysaccharide vaccine (23vPS), received 3 doses of 0.5 milliliter (mL) of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly 6 months apart and were assessed from 13vPnC Dose 3 to prior to the blood draw 28 to 42 days post-13vPnC Dose 3.
- 13vPnC (After Dose 3 Blood Draw): Participants who were previously immunized with at least 1 dose of 23-valent pneumococcal polysaccharide vaccine (23vPS), received at least 1 of the 3 doses of 0.5 milliliter (mL) of 13-valent pneumococcal conjugate vaccine (13vPnC) intramuscularly 6 months apart and were assessed from the blood draw 28 to 42 days post-13vPnC Dose 3 up to 6-month follow-up.
Arm/Group | 13vPnC (After Dose 1 and Before Dose 2) | 13vPnC (After Dose 2 and Before Dose 3) | 13vPnC (After Dose 3 and Before Dose 3 Blood Draw) | 13vPnC (After Dose 3 Blood Draw)
Serious Adverse Events (participants affected / at risk) | 24/329 | 14/300 | 4/278 | 10/329
Other Adverse Events (participants affected / at risk) | 244/329 | 196/300 | 169/278 | 30/329
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13vPnC (After Dose 1 and Before Dose 2) (N=329) | 13vPnC (After Dose 2 and Before Dose 3) (N=300) | 13vPnC (After Dose 3 and Before Dose 3 Blood Draw) (N=278) | 13vPnC (After Dose 3 Blood Draw) (N=329)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 3 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 2 | 0 | 0
Prinzmetal angina (Cardiac disorders) | 0 | 1 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Mediastinal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Mycobacterium abscessus infection (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Anal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Cytomegalovirus hepatitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 2
Carcinoma in situ of penis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Complicated migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 1 | 1
Bladder prolapse (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Aortic stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | 13vPnC (After Dose 1 and Before Dose 2) (N=329) | 13vPnC (After Dose 2 and Before Dose 3) (N=300) | 13vPnC (After Dose 3 and Before Dose 3 Blood Draw) (N=278) | 13vPnC (After Dose 3 Blood Draw) (N=329)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Polycythaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 1
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 3 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Eustachian tube disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0
Episcleritis (Eye disorders) | 0 | 0 | 0 | 1
Iritis (Eye disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 1 | 0 | 3
Oral pain (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Anogenital dysplasia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 3
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diverticulum (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 6 | 1 | 2 | 0
Fatigue (General disorders) | 4 | 8 | 1 | 1
Influenza like illness (General disorders) | 2 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 1 | 0 | 0
Injection site pain (General disorders) | 1 | 0 | 0 | 0
Injection site paraesthesia (General disorders) | 1 | 0 | 0 | 0
Oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 2 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 2 | 2 | 2 | 0
Food allergy (Immune system disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 17 | 8 | 1 | 0
Folliculitis (Infections and infestations) | 5 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 2 | 4 | 0
Laryngitis (Infections and infestations) | 3 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 3 | 1 | 3 | 0
Body tinea (Infections and infestations) | 2 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 2 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 2 | 0 | 2 | 0
Syphilis (Infections and infestations) | 2 | 1 | 0 | 0
Bronchitis viral (Infections and infestations) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 1 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Urethritis (Infections and infestations) | 1 | 1 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 3 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 2 | 1 | 0
Kidney infection (Infections and infestations) | 0 | 2 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Balanitis candida (Infections and infestations) | 0 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 1 | 2
Giardiasis (Infections and infestations) | 0 | 1 | 0 | 0
Gonorrhoea (Infections and infestations) | 0 | 1 | 0 | 0
Post viral fatigue syndrome (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 1
Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Keratitis herpetic (Infections and infestations) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Salmonellosis (Infections and infestations) | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Anal pap smear abnormal (Investigations) | 2 | 0 | 0 | 0
Prostatic specific antigen increased (Investigations) | 2 | 0 | 0 | 0
Weight increased (Investigations) | 2 | 0 | 0 | 0
Blood pressure increased (Investigations) | 1 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 1 | 1 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 1 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 0 | 0
Viral load increased (Investigations) | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 1
Tuberculin test positive (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 2
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 1 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia intercostal (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Oral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Cervicitis human papilloma virus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 9 | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 2 | 0 | 1
Migraine (Nervous system disorders) | 1 | 2 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Cervicobrachial syndrome (Nervous system disorders) | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 3 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 2 | 0 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Fear (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Substance abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Tobacco abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 2 | 0 | 0
Anxiety disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Major depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1
Genital pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Gynaecomastia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine cervical squamous metaplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Vulvar dysplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Epididymal cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 3 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 2
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 7 | 4 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Eczema nummular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 2 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 1 | 0 | 0 | 0
Redness (Any) (Skin and subcutaneous tissue disorders) | 9/162 | 10/122 | 10/105 | 0/0
Redness (Mild) (Skin and subcutaneous tissue disorders) | 7/161 | 8/120 | 9/104 | 0/0
Redness (Moderate) (Skin and subcutaneous tissue disorders) | 2/158 | 2/117 | 4/102 | 0/0
Redness (Severe) (Skin and subcutaneous tissue disorders) | 0/157 | 2/117 | 1/101 | 0/0
Swelling (Any) (Skin and subcutaneous tissue disorders) | 11/162 | 16/126 | 12/107 | 0/0
Swelling (Mild) (Skin and subcutaneous tissue disorders) | 10/161 | 15/125 | 9/106 | 0/0
Swelling (Moderate) (Skin and subcutaneous tissue disorders) | 1/158 | 1/116 | 4/102 | 0/0
Swelling (Severe) (Skin and subcutaneous tissue disorders) | 1/158 | 2/117 | 1/101 | 0/0
Pain (Any) (Skin and subcutaneous tissue disorders) | 205/260 | 193/237 | 167/204 | 0/0
Pain (Mild) (Skin and subcutaneous tissue disorders) | 197/258 | 181/230 | 158/197 | 0/0
Pain (Moderate) (Skin and subcutaneous tissue disorders) | 32/173 | 50/150 | 39/129 | 0/0
Pain (Severe) (Skin and subcutaneous tissue disorders) | 2/158 | 10/123 | 6/105 | 0/0
Fever (>=38 degrees C) (General disorders) | 10/162 | 6/117 | 8/104 | 0/0
Fever (>=38 but <38.5 degrees C) (General disorders) | 6/160 | 5/116 | 5/104 | 0/0
Fever (>=38.5 but <39 degrees C) (General disorders) | 2/157 | 1/116 | 1/101 | 0/0
Fever (>=39 but =<40 degrees C) (General disorders) | 2/159 | 0/115 | 2/101 | 0/0
Fever (>40 degrees C) (General disorders) | 1/158 | 0/115 | 0/101 | 0/0 — Report of fever >40 degrees C after 13vPnC Dose 1 was confirmed as data entry error.
Fatigue (Any) (General disorders) | 141/235 | 119/188 | 90/160 | 0/0
Fatigue (Mild) (General disorders) | 121/223 | 101/176 | 72/149 | 0/0
Fatigue (Moderate) (General disorders) | 75/200 | 59/154 | 48/132 | 0/0
Fatigue (Severe) (General disorders) | 10/163 | 9/121 | 6/105 | 0/0
Headache (Any) (General disorders) | 138/224 | 97/173 | 64/137 | 0/0
Headache (Mild) (General disorders) | 124/216 | 80/165 | 53/130 | 0/0
Headache (Moderate) (General disorders) | 57/183 | 44/142 | 29/118 | 0/0
Headache (Severe) (General disorders) | 5/160 | 4/117 | 5/103 | 0/0
Vomiting (Any) (General disorders) | 19/164 | 9/120 | 12/109 | 0/0
Vomiting (Mild) (General disorders) | 19/164 | 8/119 | 9/107 | 0/0
Vomiting (Moderate) (General disorders) | 0/157 | 1/116 | 5/104 | 0/0
Vomiting (Severe) (General disorders) | 0/157 | 0/115 | 0/101 | 0/0
Diarrhea (Any) (General disorders) | 85/193 | 69/155 | 52/134 | 0/0
Diarrhea (Mild) (General disorders) | 77/191 | 58/147 | 47/131 | 0/0
Diarrhea (Moderate) (General disorders) | 21/166 | 20/130 | 13/109 | 0/0
Diarrhea (Severe) (General disorders) | 3/160 | 6/119 | 2/103 | 0/0
New generalized muscle pain (Any) (General disorders) | 152/234 | 143/199 | 112/170 | 0/0
New generalized muscle pain (Mild) (General disorders) | 139/230 | 124/188 | 95/155 | 0/0
New generalized muscle pain (Moderate) (General disorders) | 54/183 | 59/153 | 41/132 | 0/0
New generalized muscle pain (Severe) (General disorders) | 6/161 | 13/125 | 11/110 | 0/0
New generalized joint pain (Any) (General disorders) | 69/193 | 60/150 | 41/129 | 0/0
New generalized joint pain (Mild) (General disorders) | 55/185 | 50/144 | 31/119 | 0/0
New generalized joint pain (Moderate) (General disorders) | 33/172 | 29/135 | 24/120 | 0/0
New generalized joint pain (Severe) (General disorders) | 2/159 | 4/119 | 6/106 | 0/0
Bereavement (Social circumstances) | 0 | 1 | 0 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.